CLINICAL TRIAL: NCT00844857
Title: Study to Assess the Efficacy and Safety of Olanzapine and Fluoxetine Combination Versus Placebo in Patients Ages 10-17 in the Treatment of Major Depressive Episodes Associated With Bipolar I Disorder
Brief Title: A Study for Assessing Treatment of Patients Ages 10-17 With Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12116; H6P-MC-HDAX (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Results first posted 2013-02-18 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-01

CONDITIONS: Bipolar Depression
Keywords: Bipolar I Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — olanzapine-fluoxetine combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olanzapine/Fluoxetine Combination (Experimental)
  Interventions: Drug: Olanzapine Fluoxetine Combination (OFC)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olanzapine Fluoxetine Combination (OFC) — OFC doses are capsules of 3 milligrams (mg) olanzapine and 25 mg fluoxetine (3/25), 6/25, 12/25, 6/50, or 12/50 mg to be taken orally once daily in the evening for 8 weeks.
  Other Names: LY900000; Symbyax
  Arms: Olanzapine/Fluoxetine Combination
Drug: Placebo — Orally, once daily in the evening for 8 weeks.
  Arms: Placebo

SUMMARY:
The main goal of this study is to help answer the following research question(s) and not to treat the child's illness.

* Can this study drug make children with bipolar depression feel better?
* Does this study drug work better than a placebo (sugar pill)?
* Does this study drug cause side effects in children who take it?
* Is this drug safe to use in children? (The study drug is a mixture of olanzapine and fluoxetine)

ELIGIBILITY:
Inclusion Criteria:

* Male or female inpatients or outpatients, 10-17 years of age, who have not reached their 18th birthday prior to screening. Patient must weigh at least 20 kilograms (kg) at screening.
* Must meet diagnostic criteria for current major depressive episode of Bipolar I Disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Version (DSM-IV-TR) and confirmed by Kiddie Schedule for Affective Disorders and Schizophrenia for School Aged Children-Present and Lifetime (K-SADS-PL)
* Patients entering the study will also be scored by the Children's Depression Rating Scale-Revised (CDRS-R) (entry score of greater than or equal to 40) as well as the adolescent-structured Young Mania Rating Scale (YMRS) (entry score of less than or equal to 15 with YMRS Item 1 [elevated mood] score less than equal to 2).

Exclusion Criteria:

* Patients will be excluded if they are, in the opinion of the investigator, actively suicidal
* Have an acute, serious or unstable medical condition
* Have clinically significant laboratory abnormalities
* Have had one or more seizures of unclear etiology
* Have a current or lifetime diagnosis of any of the following according to DSM-IV criteria: Schizophrenia, Schizophreniform Disorder, Schizoaffective Disorder, Delusional Disorder, Psychotic Disorder Not Otherwise Specified, Delirium of any type, Amnestic Disorder, any Substance-Induced Disorder, or any Psychotic Disorder due to a General Medical Condition, unless there is substantive reason to believe patient was misdiagnosed

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 291 (Actual)
Dates: Start 2009-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California, United States
- Russia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lipetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saratov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stavropol
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tver'
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yaroslavl

REFERENCES:
- [Derived] Walker DJ, DelBello MP, Landry J, D'Souza DN, Detke HC. Quality of life in children and adolescents with bipolar I depression treated with olanzapine/fluoxetine combination. Child Adolesc Psychiatry Ment Health. 2017 Jul 12;11:34. doi: 10.1186/s13034-017-0170-7. eCollection 2017. PMID 28706563
- [Derived] Detke HC, DelBello MP, Landry J, Usher RW. Olanzapine/Fluoxetine combination in children and adolescents with bipolar I depression: a randomized, double-blind, placebo-controlled trial. J Am Acad Child Adolesc Psychiatry. 2015 Mar;54(3):217-24. doi: 10.1016/j.jaac.2014.12.012. Epub 2014 Dec 29. PMID 25721187

RESULTS

PARTICIPANT FLOW:
Groups:
- Olanzapine/Fluoxetine Combination: Olanzapine/fluoxetine Combination (OFC) 3 milligrams (mg) olanzapine and 25 mg fluoxetine (OFC 3/25) administered orally as an initial dose beginning at randomization, 6/25 mg at Visit 3 (Day 3), 6/50 mg at Visit 4 (Week 1), and 12/50 mg at Visit 5 (Week 2). If no tolerability or safety issues occurred after Visit 5 the participant continued on the maximum tolerated dose, not to exceed 12/50 mg and not less than 6/25 mg, for a total of 8 weeks.
- Placebo: Matched placebo capsule administered orally once daily for 8 weeks.
Period: Overall Study
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Started | 194 | 97
Population Analyzed | 170 (Randomized participants who took at least 1 dose of study drug excluding 2 GCP noncompliant sites.) | 85 (randomized participants who took at least 1 dose of study drug excluding 2 GCP noncompliant sites.)
Completed | 116 | 60
Not Completed | 78 | 37
Not completed — Adverse Event | 24 | 5
Not completed — Sponsor Decision | 1 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Parent/Caregiver Decision | 6 | 2
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Protocol Violation | 6 | 0
Not completed — Lack of Efficacy | 5 | 5
Not completed — Clinical Relapse | 0 | 1
Not completed — Entry Criteria Not Met | 0 | 1
Not completed — Lost to Follow-up | 2 | 3
Not completed — Did Not Take Study Drug | 3 | 1
Not completed — Good Clinical Practice Violations | 21 | 11

BASELINE CHARACTERISTICS:
Groups:
- Olanzapine/Fluoxetine Combination: OFC 3/25 mg administered orally as an initial dose beginning at randomization, 6/25 mg at Visit 3 (Day 3), 6/50 mg at Visit 4 (Week 1), and 12/50 mg at Visit 5 (Week 2). If no tolerability or safety issues occurred after Visit 5 the participant continued on the maximum tolerated dose, not to exceed 12/50 mg and not less than 6/25 mg, for a total of 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo | Total
Number analyzed (Participants) | 170 | 85 | 255
Age Continuous [Mean (Standard Deviation); unit: years] | 14.59 (2.30) | 15.03 (2.13) | 14.74 (2.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 39 | 125
  Male | 84 | 46 | 130
Region of Enrollment [Number; unit: participants]
  United States | 123 | 65 | 188
  Russian Federation | 31 | 13 | 44
  Mexico | 16 | 7 | 23
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 38 | 23 | 61
  Not Hispanic or Latino | 132 | 61 | 193
  Missing, participant did not reply | 0 | 1 | 1
Race [Number; unit: participants]
  American Indian or Alaska Native | 9 | 5 | 14
  Asian | 0 | 0 | 0
  Black or African American | 23 | 11 | 34
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 119 | 61 | 180
  Multiple | 15 | 7 | 22
  Missing, participant did not reply | 3 | 1 | 4
Number of Previous Episodes of Mania During Participants Life [Mean (Standard Deviation); unit: episodes] | 3.91 (10.43) | 3.75 (5.69) | 3.85 (9.12)
Number of Previous Episodes of Depression During Participants Life [Mean (Standard Deviation); unit: episodes] | 4.63 (9.13) | 4.11 (6.58) | 4.45 (8.36)
Number of Previous Mixed Episodes During Participants Life [Mean (Standard Deviation); unit: episodes] — A Mixed Episode is characterized by a period of time in which the criteria are met both for a Manic Episode and for a Major Depressive Episode nearly every day.
  episodes | 1.79 (7.69) | 1.53 (3.96) | 1.70 (6.68)
Number of Previous Episodes of Mania in Past 12 Months [Mean (Standard Deviation); unit: episodes] | 1.26 (3.91) | 1.27 (1.89) | 1.27 (3.37)
Number of Previous Episodes of Depression in Past 12 Months [Mean (Standard Deviation); unit: episodes] | 1.88 (4.16) | 1.71 (2.31) | 1.82 (3.64)
Number of Previous Mixed Episodes in Past 12 Months [Mean (Standard Deviation); unit: episodes] — A Mixed Episode is characterized by a period of time in which the criteria are met both for a Manic Episode and for a Major Depressive Episode nearly every day.
  episodes | 0.68 (3.97) | 0.39 (1.05) | 0.58 (3.29)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Children's Depression Rating Scale Revised (CDRS-R) Total Score at Week 8
Description: CDRS-R Total score measures the presence and severity of depression in children. The scale consists of 17 items scored on a 1-to-5- or 1-to-7-point scale. A rating of 1 indicates normal functioning. Total scores range from 17 to 113. In general, scores below 20 indicate an absence of depression, scores of 20 to 30 indicate borderline depression, and scores of 40 to 60 indicate moderate depression. Least Square (LS) mean was adjusted for baseline, country, treatment, visit, and treatment times (*) visit interaction.
Time Frame: Baseline, Week 8
Population: Population analyzed was the Modified Intention-to-Treat (M-ITT) Population: defined as all randomized participants who took at least 1 dose of study drug and excluding participants from 2 Good Clinical Practice (GCP) noncompliant sites and who had a baseline and at least 1 post-baseline CDRS-R measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Matched placebo capsule administered orally, once daily for 8 weeks.
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 170 | 84
units on a scale | -28.43 (1.13) | -23.40 (1.49)
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; Tested was the null hypothesis that there was no difference in mean changes from baseline to Week 8 between OFC and placebo. A conservative estimate of effect size of 0.4 was used in the sample size estimation for this study. A randomized ratio of 2:1 provided a 90% power with an effect size of 0.4; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — The a priori threshold for statistical significance was 0.05. Mixed Model Repeated Measures Analysis (MMRM) terms included baseline, country, treatment, visit, and treatment * visit interaction

2. Secondary Outcome: Percentage of Participants With Remission Up to Week 8
Description: Remission is defined as a CDRS-R total score less than or equal to (≤)28, and Young Mania Rating Scale (YMRS) total score ≤ 8 and Clinical Global Impressions-Bipolar Version (CGI-BP) total score ≤3. CDRS-R is a 17-item scale measuring presence/severity of depression in children and is scored on a 1-to-5- or 1-to-7-point scale. Rating of 1 indicates normal function. Scores range: 17 to 113. Scores <20 indicate an absence of depression, scores 20 to 30 indicate borderline depression, scores 40 to 60 indicate moderate depression. The YMRS is an 11-item scale measuring severity of manic episodes; 4 items are rated on a scale from 0 (symptoms not present) to 8 (symptom extremely severe) with remaining items rated on a scale from 0 (symptoms not present) to 4 (symptom extremely severe). YMRS score ranges from 0 to 60. CGI-BP measures participant's overall severity of bipolar symptoms. Scores range: 1 (normal, not at all ill ) to 7 (among the most extremely ill participants).
Time Frame: Baseline up to Week 8
Population: Population analyzed was the M-ITT Population: all randomized participants who took at least 1 dose of study drug and excluding participants from 2 GCP noncompliant sites and who had both the CDRS-R, YMRS and CGI-BP total scores at baseline and at least 1 post-baseline measurement; Last Observation Carried Forward (LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 156 | 76
percentage of participants | 59.0 | 43.4
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; Tested was the null hypothesis that there was no difference in proportions between OFC and placebo; Test type: Superiority or Other; p = 0.035, Fisher Exact — The a priori threshold for statistical significance was 0.05

3. Secondary Outcome: Percentage of Participants With Response Up to Week 8
Description: Response is defined as a CDRS-R total score greater than or equal to (≥)50% reduction from baseline and YMRS elevated mood score ≤2. CDRS-R Total score measure the presence and severity of depression in children. The scale consists of 17 items scored on a 1-to-5- or 1-to-7-point scale. Rating of 1 indicates normal function. Scores range: 17 to 113. In general, <20 indicate an absence of depression, scores 20 to 30 indicate borderline depression, and scores of 40 to 60 indicate moderate depression. YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptoms not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptoms not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60.
Time Frame: Baseline up to Week 8
Population: Population analyzed was the M-ITT Population: all randomized participants who took at least 1 dose of study drug and excluding participants from 2 GCP noncompliant sites and who had all of CDRS-R and YMRS total scores at baseline and at least 1 post-baseline measurement; LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 156 | 76
percentage of participants | 78.2 | 59.2
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; Tested was the null hypothesis that there was no difference in proportions between OFC and placebo; Test type: Superiority or Other; p = 0.003, Fisher Exact — The a priori threshold for statistical significance was 0.05

4. Secondary Outcome: Percentage of Participants in Each Improvement Category Up to Week 8
Description: CDRS-R scores: No/low improvement is < 25 percent (%) of maximum reduction from baseline. Mild improvement: maximum reduction from baseline on CDRS-R score ≥ 25% up to <50% and YMRS elevated mood score ≤ 2. Moderate improvement: maximum reduction from baseline on CDRS-R score ≥50% and <75% and YMRS elevated mood score ≤ 2. Major improvement: maximum reduction from baseline on CDRS-R score ≥75% and YMRS elevated mood score ≤ 2. CDRS-R measures presence/severity of depression in children. Scale is 17 items scored 1-to-5- or 1-to-7. Rating of 1 indicates normal function. Scores range: 17 to 113. Scores < 20 absence of depression, scores 20 to 30 borderline depression, scores 40 to 60 indicate moderate depression. YMRS is an 11-item scale that measures severity of manic episodes. Four items rated 0 (symptoms not present) to 8 (symptom extremely severe). Remaining items rated 0 (symptoms not present) to 4 (symptom extremely severe). Score range: 0 to 60.
Time Frame: Baseline up to Week 8
Population: Population analyzed was the M-ITT Population: all randomized participants who took at least 1 dose of study drug and excluding participants from 2 GCP noncompliant sites and who had both CDRS-R and YMRS total scores with a baseline and at least 1 post-baseline measurement; LOCF.
Measure: Number; unit: percentage of participants
Groups:
- Olanzapine Plus Fluoxetine Combination: OFC 3/25 mg administered orally as an initial dose beginning at randomization, 6/25 mg at Visit 3 (Day 3), 6/50 mg at Visit 4 (Week 1), and 12/50 mg at Visit 5 (Week 2). If no tolerability or safety issues occurred after Visit 5 the participant continued on the maximum tolerated dose, not to exceed 12/50 mg and not less than 6/25 mg, for a total of 8 weeks.
Arm/Group | Olanzapine Plus Fluoxetine Combination | Placebo
Number analyzed (Participants) | 156 | 76
percentage of participants
  No or Low Improvement | 12.8 | 22.4
  Mild Improvement | 9.0 | 18.4
  Moderate Improvement | 21.8 | 18.4
  Major Improvement | 56.4 | 40.8
Statistical Analysis 1: Comparison: Olanzapine Plus Fluoxetine Combination vs Placebo; Tested was the null hypothesis that there was no difference in proportions between OFC and placebo; Test type: Superiority or Other; p = 0.007, Ordinal Logistic Regression — The a priori threshold for statistical significance was 0.05. Ordinal Logistic Regression Model terms include baseline CDRS-R, baseline YMRS, and treatment

5. Secondary Outcome: Change From Baseline in the YMRS Total Score at Week 8
Description: The YMRS is an 11-item scale measuring the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total scores ranges: 0 to 60. LS mean was adjusted for baseline, country, treatment, visit, and treatment * visit interaction.
Time Frame: Baseline, Week 8
Population: Population analyzed was the M-ITT Population: all randomized participants who took at least 1 dose of study drug and excluding participants from 2 GCP noncompliant sites who had YMRS total scores with a baseline and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 118 | 60
units on a scale | -2.02 (0.47) | -1.57 (0.63)
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; Tested was the null hypothesis that there was no difference in mean changes from baseline to Week 8 between OFC and placebo; Test type: Superiority or Other; p = 0.527, Mixed Models Analysis — The a priori threshold for statistical significance was 0.05. MMRM terms included baseline, country, treatment, visit, and treatment*visit interaction

6. Secondary Outcome: Change From Baseline in the Clinical Global Impression Scale - Bipolar Version (CGI-BP) Score at Week 8
Description: CGI-BP measures severity of illness for bipolar illness. Scores range: 1 (normal, not ill at all) to 7 (among the most extremely ill patients). LS mean was adjusted for baseline, country, treatment, visit, and treatment * visit interaction.
Time Frame: Baseline, Week 8
Population: Population analyzed was the M-ITT Population: all randomized participants who took at least 1 dose of study drug and excluding participants from 2 GCP noncompliant sites and who had CGI-BP total scores at baseline and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Olanzapine/Fluoxetine Combination: OFC 3/25 mg administered orally as an initial dose beginning at randomization, 6/25 mg at Visit 3 (Day 3), 6/50 mg at Visit 4 (Week 1), and 12/50 mg at Visit 5 (Week 2). If no tolerability or safety issues occurred after Visit 5 the participant continued on the maximum tolerated dose, not to exceed 12/50 mg and not less than 6/25, mg for a total of 8 weeks.
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 118 | 60
units on a scale | -2.21 (0.11) | -1.83 (0.15)
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

7. Secondary Outcome: Change From Baseline in the CDRS-R Total Score Up to Week 8
Description: CDRS-R Total score measure the presence and severity of depression in children and consists of 17 items scored on a 1-to-5- or 1-to-7-point scale. Rating of 1 indicates normal function. Total scores range from 17 to 113. In general, scores < 20 indicate an absence of depression, scores of 20 to 30 indicate borderline depression, and scores of 40 to 60 indicate moderate depression. LS mean was adjusted for baseline, country, and treatment.
Time Frame: Baseline, Week 8
Population: Population analyzed was the M-ITT Population: all randomized participants who took at least 1 dose of study drug and excluding participants from 2 GCP noncompliant sites who had CDRS-R total scores at baseline and at least 1 post-baseline measurement; LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 170 | 84
units on a scale | -28.57 (1.41) | -23.38 (1.75)
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; Tested was the null hypothesis that there was no difference in mean changes from baseline to up to Week 8 between OFC and placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — The a priori threshold for statistical significance was 0.05. ANCOVA (analysis of covariance) Model terms included baseline, country, and treatment

8. Secondary Outcome: Percentage of Participants With at Least One Treatment-Emergent Incident of Akathisia Up to Week 8
Description: Akathisia was measured using the Barnes Akathisia Rating Scale where the global scores range from 0 (absent) to 5 (severe) and a score ≥ 2 is considered abnormal.
Time Frame: Baseline up to Week 8
Population: Population analyzed was the M-ITT Population: all randomized participants who took at least 1 dose of study drug excluding participants from 2 GCP noncompliant sites; LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 159 | 79
percentage of participants | 1.3 | 0.0
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; Tested was the null hypothesis that there was no difference in proportions between OFC and placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact — The a priori threshold for statistical significance was 0.05

9. Secondary Outcome: Percentage of Participants With Treatment Emergent Suicidal Ideation or Behavior Up to Week 8
Description: Columbia-Suicide Severity Rating Scale (C-SSRS) captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Percentage of participants with suicidal ideation, behavior, and acts are provided. Suicidal ideation: a "yes" answer to any 1 of 5 suicidal ideation questions, which includes wish to be dead, and 4 different categories of active suicidal ideation. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal act: a "yes" answer to actual attempt or completed suicide.
Time Frame: Baseline up to Week 8
Population: Population analyzed was the M-ITT Population: all randomized participants who took at least 1 dose of study drug and excluding participants from 2 GCP noncompliant sites; LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 170 | 84
percentage of participants
  Total Suicidal Ideation (1 - 5) | 10.6 | 15.5
  Total Suicidal Behavior (6 - 10) | 1.8 | 2.4
  Total Suicidal Ideation or Behavior (1 - 10) | 10.6 | 15.5
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; Tested was the null hypothesis that there was no difference in proportions between OFC and placebo; Test type: Superiority or Other; p = 0.309, Fisher Exact — P-value for Suicidal Ideation. The a priori threshold for statistical significance was 0.05
Statistical Analysis 2: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; Tested was the null hypothesis that there was no difference in proportions between OFC and placebo; Test type: Superiority or Other; p = 0.667, Fisher Exact — P-value for Suicidal Behavior. The a priori threshold for statistical significance was 0.05
Statistical Analysis 3: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; Tested was the null hypothesis that there was no difference in proportions between OFC and placebo; Test type: Superiority or Other; p = 0.309, Fisher Exact — P-value for Suicidal Ideation or Behavior. The a priori threshold for statistical significance was 0.05

10. Secondary Outcome: Percentage of Participants With at Least One Incident of Worsening of Mania Up to Week 8
Description: Worsening of mania was defined as YMRS score of ≥20 and a CGI severity of mania score of ≥ 5 at the same visit. The YMRS is an 11-item scale measuring severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe) with remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60. CGI measures severity of the participant's overall severity of bipolar symptoms and scores range from 1 (normal) to 7 (among the most extremely ill participants).
Time Frame: Baseline up to Week 8
Population: Population analyzed was the M-ITT Population: all randomized participants who took at least 1 dose of study drug and excluding participants from 2 GCP noncompliant sites with YMRS and CGI total scores at baseline and at least 1 post-baseline measurement; LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 170 | 84
percentage of participants | 1.2 | 0.0
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; Tested was the null hypothesis that there was no difference in proportions between OFC and placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact — The a priori threshold for statistical significance was 0.05

11. Secondary Outcome: Change From Baseline in Symptoms of Attention-Deficit/Hyperactivity Disorder Up to Week 8
Description: Attention Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version (ADHDRS-IV-PI): Investigator Administered and Scored measures the 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Scores range: 0 to 54. The LS mean was adjusted for baseline and treatment.
Time Frame: Baseline up to Week 8
Population: Population analyzed was the M-ITT Population: all randomized participants who took at least 1 dose of study drug and excluding participants from 2 GCP noncompliant sites and ADHDRS-IV-PI results at baseline and at least 1 post-baseline measurement; LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 152 | 74
units on a scale | -4.31 (0.70) | -3.57 (1.00)
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.545, ANCOVA — P-value for ADHDRS-IV-PI Total Score. The a priori threshold for statistical significance was 0.05. ANCOVA Model terms included baseline, country and treatment

12. Secondary Outcome: Change From Baseline in the Quality of Life Questionnaire for Children and Adolescents (KINDL) Parent Scale Up to Week 8
Description: The KINDL consists of 24 Likert-scale items. Total scores were standardized to a 0 (lowest quality of life) to 100 (highest quality of life). LS mean was adjusted for baseline, country, and treatment.
Time Frame: Baseline, Week 8
Population: Population analyzed was the M-ITT Population: all randomized participants who took at least 1 dose of study drug and excluding participants from 2 GCP noncompliant sites and KINDL Parent Scale at baseline and at least 1 post-baseline measurement; LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 83 | 39
units on a scale | 15.98 (1.94) | 10.88 (2.56)
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.066, ANCOVA — The a priori threshold for statistical significance was 0.05. ANCOVA Model terms included baseline, country and treatment

13. Other Pre Specified Outcome: Percentage of Participants With at Least One Treatment-Emergent Incident of Parkinsonism Up to Week 8
Description: Parkinsonism was measured using the Simpson-Angus Scale with a total scores range from 0 to 40. A score > 3 was considered abnormal. Simpson-Angus Scale consists of 10 items, each rated on a 5-point scale, 0 (complete absence of the condition) to 4 (presence of the condition in extreme form).
Time Frame: Baseline, Week 8
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 158 | 80
percentage of participants | 0.6 | 1.3
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; Tested was the null hypothesis that there was no difference in proportions between OFC and placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact — The a priori threshold for statistical significance was 0.05

14. Other Pre Specified Outcome: Percentage of Participants With at Least One Treatment-Emergent Incident of Dyskinesia Up to Week 8
Description: Dyskinesia was measured using the Abnormal Involuntary Movement Scale (AIMS) a 12-item scale designed to record the occurrence of dyskinetic movements. Items 1 through 10 are rated on a 5-point scale: 0 (no dyskinetic movements) to 4 (severe dyskinetic movements). Items 11 and 12 are yes/no questions regarding the dental condition of a patient. Total score (0-40) is obtained by adding the scores of the first 10 items. An abnormal result is defined as having a score ≥3 for at least 1 of the first 7 items or a score ≥2 for at least two of the first 7 items.
Time Frame: Baseline, Week 8
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 160 | 80
percentage of participants | 0.6 | 0.0
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; Tested was the null hypothesis that there was no difference in proportions between OFC and placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact — The a priori threshold for statistical significance was 0.05

15. Other Pre Specified Outcome: Change From Baseline in the Quality of Life Questionnaire for Children and Adolescents (KINDL) Kid and Kiddo Combined Scale Up to Week 8
Description: The KINDL consists of 24 Likert-scale items. Kid-KINDL was administered to ages 8-11 and Kiddo-KINDL to ages 12-16. Total scores were standardized to a 0 (lowest quality of life) to 100 (highest quality of life). LS mean was adjusted for baseline, country, and treatment.
Time Frame: Baseline, Week 8
Population: Population analyzed was the M-ITT Population: all randomized participants who took at least 1 dose of study drug excluding participants from 2 GCP noncompliant sites and had KINDL Kid and Kiddo results at baseline and at least 1 post-baseline measurement. Due to small number of 10- and 11-year olds results from the 2 versions were pooled; LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 107 | 40
units on a scale | 12.83 (1.65) | 7.91 (2.40)
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.050, ANCOVA — [p-value comment as in outcome 12, analysis 1]

16. Other Pre Specified Outcome: Change From Baseline in Weight Up to Week 8
Description: Weight LS mean was adjusted for baseline and treatment.
Time Frame: Baseline, Week 8
Population: Population analyzed was the M-ITT Population: all randomized participants who took at least 1 dose of study drug and excluding participants from 2 GCP noncompliant sites and weight at baseline and at least 1 post-baseline measurement; LOCF.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 170 | 84
kilogram (kg) | 4.37 (0.23) | 0.50 (0.33)
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The a priori threshold for statistical significance was 0.05. ANCOVA Model terms included baseline and treatment

17. Other Pre Specified Outcome: Change From Baseline in Fasting Metabolic Parameters Up to Week 8
Description: Fasting glucose, fasting cholesterol and fasting triglycerides. LS means were adjusted for baseline and treatment.
Time Frame: Baseline, Week 8
Population: Population analyzed was the M-ITT Population: all randomized participants who took at least 1 dose of study drug excluding participants from 2 GCP noncompliant sites and fasting glucose, cholesterol and triglycerides at baseline and at least 1 post-baseline measurement; LOCF.
Measure: Least Squares Mean (Standard Error); unit: millimoles/liter (mmol/L)
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 158 | 81
millimoles/liter (mmol/L)
  Fasting Glucose (157, 79) | 0.03 (0.04) | 0.03 (0.06)
  Fasting Cholesterol (158, 81) | 0.42 (0.05) | -0.11 (0.07)
  Fasting Triglycerides (158, 81) | 0.40 (0.06) | -0.04 (0.08)
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.980, ANCOVA — P-value for Fasting Glucose. The a priori threshold for statistical significance was 0.05. ANCOVA Model terms included baseline and treatment
Statistical Analysis 2: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Fasting Cholesterol. The a priori threshold for statistical significance was 0.05. ANCOVA Model terms included baseline and treatment
Statistical Analysis 3: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Fasting Triglycerides. The a priori threshold for statistical significance was 0.05. ANCOVA Model terms included baseline and treatment

18. Other Pre Specified Outcome: Change From Baseline in Alanine Aminotransferase/Serum Glutamic-Pyruvic Transaminase (ALT/SGPT) Up to Week 8
Description: ALT/SGPT LS mean was adjusted for baseline and treatment.
Time Frame: Baseline, Week 8
Population: Population analyzed was the M-ITT Population: all randomized participants who took at least 1 dose of study drug and excluding participants from 2 GCP noncompliant sites and ALT/SGPT at baseline and at least 1 post-baseline measurement; LOCF.
Measure: Least Squares Mean (Standard Deviation); unit: units/Liter (U/L)
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 170 | 84
units/Liter (U/L) | 7.63 (1.46) | 0.46 (2.08)
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.005, ANCOVA — The a priori threshold for statistical significance was 0.05. ANCOVA Model terms included baseline and treatment

19. Other Pre Specified Outcome: Change From Baseline in Prolactin Up to Week 8
Description: Prolactin LS mean was adjusted for baseline and treatment.
Time Frame: Baseline, Week 8
Population: Population analyzed was the M-ITT Population: all randomized participants who took at least 1 dose of study drug and excluding participants from 2 GCP noncompliant sites and prolactin at baseline and at least 1 post-baseline measurement; LOCF.
Measure: Least Squares Mean (Standard Error); unit: microgram/Liter (μg/L)
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 170 | 84
microgram/Liter (μg/L) | 8.66 (0.77) | 0.70 (1.10)
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The a priori threshold for statistical significance was 0.05. ANCOVA Model terms included baseline and treatment

20. Other Pre Specified Outcome: Change From Baseline in Electrocardiogram (ECG) QTcF Interval Up to Week 8
Description: QTcF is defined as ECG QT interval corrected for heart rate using the Fridericia correction factor.
Time Frame: Baseline, Week 8
Population: Population analyzed M-ITT Population: all randomized participants who took at least 1 dose of study drug and excluding participants from 2 GCP noncompliant sites and QTcF at baseline and at least 1 post-baseline measurement; LOCF.
Measure: Least Squares Mean (Standard Error); unit: millisecond (msec)
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Number analyzed (Participants) | 158 | 78
millisecond (msec) | 8.19 (1.01) | -1.07 (1.44)
Statistical Analysis 1: Comparison: Olanzapine/Fluoxetine Combination vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The a priori threshold for statistical significance was 0.05. ANCOVA Model terms included baseline and treatment

ADVERSE EVENTS:
Description: Adverse events were reported for all randomized participants who took at least 1 dose of study drug, excluding 2 GCP noncompliant sites.
Arm/Group | Olanzapine/Fluoxetine Combination | Placebo
Serious Adverse Events (participants affected / at risk) | 9/170 | 6/85
Other Adverse Events (participants affected / at risk) | 125/170 | 49/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Olanzapine/Fluoxetine Combination (N=170) | Placebo (N=85)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1)
Aggression aggravated (Psychiatric disorders) | 2 (3) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar affective disorder aggravated (Psychiatric disorders) | 1 (1) | 0 (0)
Depression worsened (Psychiatric disorders) | 0 (0) | 1 (1)
Homicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Psychosis aggravated (Psychiatric disorders) | 0 (0) | 1 (1)
Self injurious behavior (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (2) | 0 (0)
Ovulation disorder (Reproductive system and breast disorders) | 1/86 (1) | 0/39 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine/Fluoxetine Combination (N=170) | Placebo (N=85)
Nausea (Gastrointestinal disorders) | 8 (8) | 11 (13)
Vomiting (Gastrointestinal disorders) | 8 (8) | 5 (5)
Triglyceride increased (Investigations) | 9 (10) | 1 (1)
Weight gain (Investigations) | 32 (32) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 5 (6)
Increased appetite (Metabolism and nutrition disorders) | 28 (28) | 1 (1)
Drowsiness (Nervous system disorders) | 9 (9) | 0 (0)
Headache (Nervous system disorders) | 24 (33) | 12 (16)
Sedation (Nervous system disorders) | 11 (12) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days